CLINICAL TRIAL: NCT02232542
Title: Tolerability and Safety of 40 mg and 100 mg Duloxetine BID Given Over 7 Days in Healthy Female Subjects. A Randomised, Placebo-controlled Double-blind Trial.
Brief Title: Tolerability and Safety of Duloxetine BID in Healthy Female Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1208.1
Record Dates: First submitted 2014-09-04; First posted 2014-09-05 (Estimated); Last update posted 2014-09-05 (Estimated); Status verified 2014-08

CONDITIONS: Healthy
MeSH Terms: interventions — Duloxetine Hydrochloride

ARMS (3):
- Duloxetine - low dose (Experimental)
  Interventions: Drug: Duloxetine - low dose
- Duloxetine - high dose (Experimental)
  Interventions: Drug: Duloxetine - high dose
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine - low dose
  Arms: Duloxetine - low dose
Drug: Duloxetine - high dose
  Arms: Duloxetine - high dose
Drug: Placebo
  Arms: Placebo

SUMMARY:
Study to assess the safety and tolerability of 100 mg of duloxetine BID compared to 40 mg of duloxetine BID or placebo for 7 days

ELIGIBILITY:
Inclusion Criteria:

* Healthy female subjects as determined by results of screening
* Signed written informed consent in accordance with Good Clinical Practice (GCP) and local legislation
* Age ≥ 40 years
* BMI ≥ 18.5 and ≤ 29.9 kg/m2

Exclusion Criteria:

* Any finding at any of the medical examinations (including blood pressure, pulse rate and ECG (electrocardiogram)) deviating from normal and of clinical relevance (resting heart rate greater than 100 bpm or tachyarrhythmia)
* History of or current gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunologic, hormonal disorders (except thyroid hormones and hormonal replacement therapy)
* History of relevant orthostatic hypotension, fainting spells and blackouts
* Diseases of the central nervous system (such as epilepsy) or psychiatric disorders
* Chronic or relevant acute infections
* History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator, any bleeding disorder including prolonged or habitual bleeding, other hematologic disease, cerebral bleeding (e.g. after a car accident), commotio cerebri
* Intake of drugs with a long half-life (> 24 hours) within 1 month prior to administration
* Use of any drugs that might influence the results of the trial (especially CYP2D6 or CYP1A2 modulating substances) within 2 weeks prior to administration or during the trial
* Participation in another trial with an investigational drug within 2 months prior to administration or during trial
* Smoker (> 10 cigarettes or 3 cigars or 3 pipes/day) or inability to refrain from smoking on study days
* Alcohol abuse (> 60 g/day)
* Caffeine abuse (> 4 cups/day)
* Drug abuse
* Blood donation within 1 month prior to administration or during the trial
* Excessive physical activities within 10 days prior to administration or during the trial
* Any laboratory value outside the clinically accepted reference range
* Ineffective contraception

Min Age: 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2003-06; Primary Completion 2003-08 (Actual)

PRIMARY OUTCOMES:
Assessment of tolerability by investigator on a 4-point scale | Up to day 14 after drug administration
Number of subjects with adverse events | Up to day 14 after drug administration
Number of subjects with clinically relevant findings in electrocardiogram (ECG) | Up to day 14 after drug administration
Number of subjects with clinically relevant findings in vital signs | Up to day 14 after drug administration
  systolic and diastolic blood pressure
Number of subjects with abnormal changes in laboratory parameters | Up to day 14 after drug administration